CLINICAL TRIAL: NCT02820688
Title: Impact of Local Anesthetic Concentration-Volume Modifications on Ultrasound Guided Infraclavicular Nerve Block Effectiveness
Brief Title: Concentration-Volume Relationship in Infraclavicular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANES-IK-0609
Record Dates: First submitted 2016-06-10; First posted 2016-07-01 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Brachial Plexus Blockade
Keywords: Local Anesthtetics; Nerve Block; Bupivacaine; Prilocaine
MeSH Terms: interventions — Bupivacaine; Prilocaine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Concentrated (Active Comparator): Infraclavicular nerve block under guidance of ultrasonography will be performed using an undiluted solution of 45mg bupivacaine and 180mg prilocaine (bupivacaine 0.25% and prilocaine 1%, 18mL in total) to patients in this group
  Interventions: Drug: Bupivacaine 0.25%; Drug: Prilocaine 1%; Procedure: Infraclavicular Nerve Block; Device: Ultrasound
- Diluted by 33% (Active Comparator): Infraclavicular nerve block under guidance of ultrasonography will be performed using a solution of 45mg bupivacaine and 180mg prilocaine diluted by 33% (bupivacaine 0.167% and prilocaine 0.66%, 27mL in total) to patients in this group
  Interventions: Procedure: Infraclavicular Nerve Block; Drug: Bupivacaine 0.167%; Drug: Prilocaine 0.66%; Device: Ultrasound
- Diluted by 50% (Active Comparator): Infraclavicular nerve block under guidance of ultrasonography will be performed using a solution of 45mg bupivacaine and 180mg prilocaine diluted by 50% (bupivacaine 0.125% and prilocaine 0.5%, 36mL in total) to patients in this group
  Interventions: Procedure: Infraclavicular Nerve Block; Drug: Bupivacaine 0.125%; Drug: Prilocaine 0.5%; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacaine 0.25%
  Other Names: Marcaine
  Arms: Concentrated
Drug: Prilocaine 1%
  Other Names: Citanest
  Arms: Concentrated
Procedure: Infraclavicular Nerve Block — Ultrasound guided infraclavicular nerve block
Drug: Bupivacaine 0.167%
  Other Names: Marcaine
  Arms: Diluted by 33%
Drug: Bupivacaine 0.125%
  Other Names: Marcaine
  Arms: Diluted by 50%
Drug: Prilocaine 0.66%
  Other Names: Citanest
  Arms: Diluted by 33%
Drug: Prilocaine 0.5%
  Other Names: Citanest
  Arms: Diluted by 50%
Device: Ultrasound — All nerve blocks will be performed with ultrasound guidance

SUMMARY:
This prospective, randomized, double blind study aims to determine the optimal volume for adequate sensorial and motor blockade following an infraclavicular block. Patients will be randomized into three groups. Using a constant dose of local anesthetics (45mg bupivacaine 180mg prilocaine), different volumes will be used in each of the groups (First group; 18mL, second group; 27mL, third group; 36mL). Onset, duration and quality of sensory and motor block will be compared for patients between groups

DETAILED DESCRIPTION:
Although ultrasound guided infraclavicular nerve block is routinely used to provide anesthesia for almost all of the upper extremity surgeries, optimal volume and concentration of locak anesthetic to be administered is still a subject of debate. This prospective, randomized, double blind study aims to determine the optimal volume for adequate sensorial and motor blockade following an infraclavicular block. Patients will be randomly allocated into three groups. 81 patients (27 in each group) are planned to be enrolled in this study due to a power analysis performed (G-power ver 3.1). Using a constant dose of local anesthetics (45mg bupivacaine 180mg prilocaine), different volumes will be used in each of the groups (First group; 18mL, second group; 27mL, third group; 36mL). Onset, duration and quality of sensory and motor block will be compared for patients between groups Researchers who perform the block and assess the block quality and onset will be blinded to patients' groups. Patients will also be blinded to groups they are assigned.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for upper extremity surgery with infraclavicular nerve block

Exclusion Criteria:

* Patient Refusal
* Patients younger than 18
* Patients with known local anesthetic allergies
* Patients with a BMI>30
* Diabetic Patients
* Uncooperated Patients
* Patients with coagulopathy or recieving anticoagulant therapy
* Skin infection on injection site
* Patients diagnosed with sepsis or bacteremia
* Physiologic and emotional lability
* Surgeries that are expected to last longer than 3 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Sensory Block, as assessed by hollman scale for pinprick test | 0, 3rd, 6th, 9th, 12th, 20th, 25th, 30th minute
  Sensorial response to pinprick will be assessed at innervation sites of ulnar median radial and musculocutaneous nerves. Innervation sites of assessment are volar skin of the fifth finger for ulnar nerve, volar skin of second finger for median nerve and dorsal, proximal of the second finger for radial nerve and skin of the anterolateral forearm for musculocutaneous nerve.
Motor Block, as assessed by hollman scale for motor blockade | 0, 3rd, 6th, 9th, 12th, 20th, 25th, 30th minute
  Motor function for each nerve will be assessed. Movements to be evaluated are; abduction of the fingers for ulnar nerve, thumb opposition for median nerve, extension of the forearm for radial nerve and flexion of the forearm for musculocutaneous nerve.
Postoperative Sensory Block, as assessed by hollman scale for pinprick test | 1th hour in PACU
Postoperative Motor Block, as assessed by hollman scale for motor blockadet | 1th hour in PACU

SECONDARY OUTCOMES:
Pain, as assessed by visual analogue scale | 1st hour and 6th hour
  In addition, patients' first complaint time of pain will be recorded by nurse

CONTACTS AND LOCATIONS:
Overall Officials: Zeki T Tekgul, MD, Principal Investigator — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosaffa F, Gharaei B, Qoreishi M, Razavi S, Safari F, Fathi M, Mohseni G, Elyasi H, Hosseini F. Do the Concentration and Volume of Local Anesthetics Affect the Onset and Success of Infraclavicular Anesthesia? Anesth Pain Med. 2015 Aug 22;5(4):e23963. doi: 10.5812/aapm.23963v2. eCollection 2015 Aug. PMID 26473102
- [Background] Gonzalez AP, Bernucci F, Techasuk W, Pham K, Finlayson RJ, Tran DQ. A randomized comparison between 3 combinations of volume and concentration of lidocaine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2013 May-Jun;38(3):206-11. doi: 10.1097/AAP.0b013e318287fe53. PMID 23518863
- [Background] Fenten MG, Schoenmakers KP, Heesterbeek PJ, Scheffer GJ, Stienstra R. Effect of local anesthetic concentration, dose and volume on the duration of single-injection ultrasound-guided axillary brachial plexus block with mepivacaine: a randomized controlled trial. BMC Anesthesiol. 2015 Sep 30;15:130. doi: 10.1186/s12871-015-0110-0. PMID 26423050